CLINICAL TRIAL: NCT04687111
Title: A Randomised, Controlled, Double-blind, Double-dummy, Clinical Trial Comparing Sacubitril-Valsartan Versus Valsartan in Asymptomatic, Stage A/B HFpEF Patients With Elevated Natriuretic Peptide and Abnormal LAVI. (Previously NCT02682719)
Brief Title: Personalised Prospective Comparison of ARni With ArB in Patients With Natriuretic Peptide eLEvation
Acronym: PARABLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mark Ledwidge (Other)
Collaborators: The Heartbeat Trust (Other)
Responsible Party: Sponsor-Investigator, Mark Ledwidge, Research Director, STOP-HF Unit, St Vincent's University Hospital, Ireland
Organization: St Vincent's University Hospital, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBT-PTCL-01, SVUH-2015-002; 2015-002928-53 (EudraCT Number); NCT02682719 (obsolete NCT alias)
Record Dates: First submitted 2018-07-25; First posted 2020-12-29 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Atrial Remodeling; Myocardial Dysfunction; Left Ventricular Remodeling; Left Ventricular Diastolic Dysfunction; Hypertension; Cardiovascular Morbidity; Fibrosis Myocardial; Inflammatory Myopathy; Atrial Arrhythmia
Keywords: Natriuretic peptide; Atrial remodelling; Atrial cardiomyopathy; Asymptomatic left ventricular diastolic dysfunction; Preserved ejection fraction; Myocardial fibrosis; Myocardial inflammation; Ventricular dysfunction
MeSH Terms: conditions — Atrial Remodeling; Ventricular Remodeling; Ventricular Dysfunction, Left; Hypertension; Myositis; Myocarditis; Ventricular Dysfunction | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: Randomised, prospective, active comparator, double blind, double dummy, controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Valsartan 40mg bid titrated to maximum dose of 160mg bid
  Interventions: Drug: Valsartan
- Intervention (Experimental): Sacubitril/Valsartan 50mg bid titrated to maximum dose of 200mg bid
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Sacubitril-Valsartan is an Angiotensin Receptor blocker and Neprilysin Inhibitor
  Other Names: LCZ696; Entresto
  Arms: Intervention
Drug: Valsartan — Valsartan is an Angiotensin Receptor Blocker
  Arms: Control

SUMMARY:
Sacubitril-valsartan, an Angiotensin Receptor Blocker-Neprilysin Inhibitor (ARNI), currently marketed for the management of heart failure, has been shown to reduce cardiovascular morbidity and mortality in stage C heart failure with reduced ejection fraction. In stage C HFpEF, sacubitril-valsartan has also been shown to reduce left atrial volume index measured using echocardiography over a 9 month timeframe. The PARABLE study investigates the hypothesis that sacubitril-valsartan can provide benefits in terms of left atrial structure and function as well as left ventricular structure and function in asymptomatic (stage A/B HFpEF) patients. This is a prospective, randomised, double-blind, double-dummy, phase II study design. The patient population will have hypertension and/or diabetes together with preserved ejection fraction, elevated natriuretic peptide (NP) and abnormal left atrial volume index (LAVI, > 28 mL/m2).

DETAILED DESCRIPTION:
Background.

An effective prevention strategy is critical if the established epidemic of heart failure and cardiovascular disease is to be curbed. This is particularly important in the context of increasing community prevalence of stage B HFpEF and left ventricular diastolic abnormalities associated with hypertension and diabetes and requires community diagnostics and targeted preventative therapies. Individualising risk beyond the presence of established risk factors can be achieved with NP assessment. Elevated NP in a population with established cardiovascular disease defines a group more prone to cardiac dysfunction, heart failure and other cardiovascular events. This can be used to risk stratify asymptomatic populations, targeting those most likely to need intensive intervention and follow-up.

In the prospective, randomised, pragmatic St Vincent's Screening TO Prevent Heart Failure (STOP-HF) trial [Ledwidge 2013], NP-based screening and collaborative care with general practice provided a multi-faceted intervention for patients with risk factors for heart failure. This involved community NP screening, improved use of RAAS modifying therapy, collaborative care with general practice as well as cardiovascular coaching for patients with mild elevations of BNP (>50 pg/mL).The intervention reduced stage B and C heart failure, most of which was preserved ejection fraction, as well as major adverse cardiovascular events requiring hospitalisation. This first of type study, along with a second study in diabetes [Huelsmann 2013], indicates that a biomarker driven strategy based on NP screening amongst stage AB heart failure patients is feasible and has an impact on heart failure and other cardiovascular diseases. These studies have been incorporated into 2017 American Heart Association/American College of Cardiology guidelines as well as other international guideline recommendations in heart failure.

However, while successful, the STOP-HF biomarker strategy lacks a specific pharmacological intervention linked to the screening biomarker, NP. An analysis of the STOP-HF follow-up study, supports other work showing that the minor C allele of genetic variant rs198389 of the NPPB gene (in the promoter region) is associated with sustained, elevated circulating levels of BNP and reduced incidence of left ventricular dysfunction over a five-year follow up period. These data support the hypothesis that use of LCZ696 to pharmacologically raise NP could provide cardioprotection in stage A/B heart failure patients. As neprilysin degrades biologically active NP, LCZ696 increases myocardial cyclic guanosine monophosphate (cGMP) which reduces vascular and myocardial stiffness as well as hypertrophy. This could improve cardiac structure and performance. NPs also stimulate natriuresis, diuresis, vasodilation and have been shown to have anti-fibrotic and anti-sympathetic benefits, which could augment the STOP-HF preventative strategy with a specific pharmacological intervention. [Ledwidge 2103, Phelan 2012, Potter 2006, Gardiner 2007]. Atrial tissue gene expression of BNP in patients with stage B HFpEF is associated with atrial fibrosis, procollagen expression and presence of M2 monocyte-derived-macrophage marker CD163 [Watson 2020]. Further analyses of the STOP-HF follow-up study shows that BNP strongly associates with the presence of atrial cardiomyopathy, an independent predictor of new onset major adverse cardiovascular events.

Taken together, these data could support a role for sacubitril-valsartan versus valsartan alone in favourably modulating vascular compliance, cardiac structure, cardiac function as well as progression of left atrial structural and functional abnormalities amongst patients with stage B HFpEF. If left atrial structure and function is also associated with new onset major adverse cardiovascular events, the intervention could also modulate cardiovascular events. Finally, new CMRI imaging measures of cardiac function, such as CMR e' have been developed and will allow full characterisation of the cardiovascular impact of the intervention, including in subsets of patients with established atrial cardiomyopathy.

Rationale for the study

Elevated NP in an at-risk population independently identifies cardiovascular risk, which can be specifically targeted by LCZ696. In a small proportion of patients (<5%) with cardiovascular risk factors and elevated NP, significant asymptomatic LV systolic dysfunction will be present and for these RAAS modifying therapy is mandated. However, there is a larger group of patients with elevated NP who have stage B HFpEF, with or without diastolic dysfunction. These patients may have preclinical, or asymptomatic, left ventricular diastolic dysfunction (ALVDD), atrial cardiomyopathy (AC) or both and are at heightened risk for heart failure and other cardiovascular events [Watson 2020].

The increase in NP in stage B HFpEF, ALVDD and AC is likely a fibro-inflammatory signal, which in-turn contributes to tissue remodelling, vascular disease, myocardial stiffening and left ventricular dysfunction. For example, hypertension, a common risk factor for ALVDD, is associated with an adverse accumulation of fibrous tissue and studies have demonstrated a strong relationship between ventricular stiffness, myocardial collagen content and plasma levels of myocardial collagen turnover markers [Hogg 2004, Querejeta 2004]. Cardiac inflammation, fibrosis and hypertrophy drive the pathophysiology [Gardiner 2007, Martos 2007] associated with vascular disease, myocardial stiffening, and left atrial as well as left ventricular dysfunction. [Phelan 2012, Jannuzzi 2019] Interrupting this pathophysiological process at an early stage before the development of ventricular dysfunction may prevent or slow development to heart failure and also have an impact on the development of other cardiovascular events driven by this pathophysiological process. This may be particularly important for prevention of the development of a sub-type of stage C HFpEF characterised by older age, elevated LAVI, atrial fibrillation and chronic kidney disease, which puts patients at very high risk adverse outcome [Shah 2015]. Importantly, there is currently no specific disease modifying therapy for these patients, beyond conventional risk factor control.

Accordingly, suppressing the RAAS will reduce the pro-fibrotic impact of angiotensin II. Addition of sacubitril, which reduces degradation of endogenous, cardio-protective NPs, could reduce pulse pressure, myocardial stiffness and augment the beneficial anti-inflammatory and anti-fibrotic effects of NPs beyond conventional RAAS modifying therapy. The latter may be mediated through impacts on the innate immune system, fibro-inflammation and monocyte-derived-macrophages in the myocardium [Watson 2020].

Several studies have shown that the interplay between the myocardium and extracellular matrix (ECM) can now be evaluated via analysis of serum samples of markers of collagen turnover. [Martos 2007, Querejeta 2007] Altered serum levels of collagen markers (e.g. Collagen 1A1) and matrix metalloproteinase (e.g. MMP-2 and MMP-9) suggest increased collagen turnover associated with fibrosis in diastolic heart failure. [Martos, 2007, Ahmed 2006, Nikishimi 2006] Other biomarkers of cardiac structure and function of relevance in ALVDD/AC include Galectin 3 and ST-2, biomarkers of cardiac remodelling and tissue fibrosis. Finally, cGMP, which blunts activation pathways and diminishes hypertrophy, fibrosis, cellular toxicity, and maladaptive remodelling in the myocardium, may also be modulated by sacubitril-valsartan, not only through inhibition of breakdown of BNP, but also ANP and other vasoactive peptides [Ibrahim 2019].

In high risk patients with preserved ejection fraction, elevated LAVI reflects increased left ventricular filling pressures, fibro-inflammation and is a strong, continuous marker of diastolic dysfunction as well as future cardiovascular events. Interventions that could improve myocardial performance and reduce progression of LAVI and other structural abnormalities might also help prevent cardiac morbidity and progression to stage B/C HFpEF. Sacubitril-valsartan has been shown to modulate NP activity and reduce LAVI in comparison with valsartan in the PARAMOUNT study [Solomon 2012]. The reduction of 2.6 mL/m2 with LCZ696 compared with an increase of 0.3 mL/m2 with valsartan (p=0.007 for difference) from a baseline of 36 mL/m2 over 36 weeks appears to be clinically significant in these patients with preserved ejection fraction. However, further work is required to understand the implications of this result in stage A/B HFpEF, especially using more precisely defined myocardial structure and function with cardiac magnetic resonance imaging (cMRI). Furthermore, in the PARAGON-HF study (Solomon 2019), there was no significant benefit of sacubitril-valsartan in patients with HFpEF with respect to the primary composite outcome of hospitalisation and death. The differential effect of sacubitril-valsartan versus valsartan in relation to left ventricular ejection fraction as well as stage B versus C HFpEF requires further evaluation. No study has evaluated sacubitril-valsartan in patients with stage A/B HFpEF, elevated natriuretic peptides and abnormal LAVI.

Aim

The main aim of the PARABLE trial is to assess the impact of sacubitril-valsartan versus valsartan alone on structural, functional and biochemical abnormalities of the myocardium in an asymptomatic cohort with preserved ejection fraction, cardiovascular risk factors, abnormal LAVI and elevated NP (brain type natriuretic peptide [BNP] and/or N-terminal of the prohormone BNP [NT-proBNP]).

PARABLE tests the hypothesis that sacubitril-valsartan versus valsartan alone would result in beneficial effects on atrial and ventricular structure and function, thereby preventing progression of cardiac abnormalities in stage B HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40yrs with cardiovascular risk factor(s) including at least one of:

   1. History of hypertension (medicated for greater than one month);
   2. History of diabetes;
2. Elevated NP: Elevated NP: BNP between 20 and 280pg/ml or NT-proBNP values between 100 pg/ml and 1,000 pg/ml within 6 months prior to screening or at screening
3. LAVI > 28 mL/m2 obtained during Doppler Echocardiography within 6 months prior to screening or at screening
4. Subjects must give written informed consent to participate in the study and before any study related assessments are performed.

Exclusion Criteria:

1. A history of heart failure.
2. Asymptomatic left ventricular systolic dysfunction defined as LVEF <50% on most recent measurement.
3. Systolic blood pressure <100mmHg
4. Persistent atrial fibrillation.
5. History of hypersensitivity, allergy or intolerance to LCZ696, ARB or neprilysin therapy or to any of the excipients or other contraindication to their use.
6. Previous history of intolerance to recommended target doses for ARBs
7. Subjects who require treatment with both an ACE inhibitor and an ARB
8. Presence of haemodynamically significant mitral and /or aortic valve disease.
9. Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic stenosis.
10. Conditions that are expected to compromise survival over the study period.
11. Serum potassium level > 5.2 mmol/L at screening.
12. Severe renal insufficiency (eGFR <30 mL per minute per 1.73 m2).
13. Hepatic dysfunction (Any LFT > 3 times the upper limit of normal (ULN))
14. Concomitant use of aliskiren
15. History of angioedema.
16. History or evidence of drug or alcohol abuse within the last 12 months
17. Malignancy or presence of any other disease with a life expectancy of < 2 years
18. Women who are pregnant, breast-feeding, or women of child bearing potential not using estro-progestative oral or intra-uterine contraception or implants, or women using estro-progestative oral or intra-uterine contraception or implants but who consider stopping it during the planned duration of the study. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. (Contraception must be continued for one week following discontinuation of study drug).
19. Concomitant participation in other intervention trials
20. Participation in any investigational drug trial within one month of visit 1.
21. Refusal to provide informed consent
22. Subjects with contraindications to MRI

    1. Brain aneurysm clip
    2. Implanted neural stimulator
    3. Implanted cardiac pacemaker or defibrillator
    4. Cochlear implant
    5. Ocular foreign body (e.g. metal shavings)
    6. Other implanted medical devices: (e.g. Swan-Ganz catheter)
    7. Insulin pump
    8. Metal shrapnel or bullet.
23. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs, including but not limited to any of the following:

    1. History of major gastrointestinal tract surgery including gastrectomy, gastroenterostomy, or bowel resection.
    2. Inflammatory bowel disease during the 12 months prior to Visit 1.
    3. Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase.
    4. Evidence of hepatic disease as determined by any one of the following: SGOT or SGPT values exceeding 3 x ULN at Visit 1, a history of hepatic encephalopathy, a history of oesophageal varices, or a history of portocaval shunt.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2021-06-11 (Estimated); Study Completion 2021-06-11 (Estimated)

PRIMARY OUTCOMES:
Change in Left Atrial Volume Index (LAV/BSA*) | Baseline-18 months
  Measured as left atrial volume (Simpson's method, using a stack of short axis slices across the entire left atrium) indexed to body surface area (*DuBois formula) using Cardiac Magnetic Resonance Imaging (cardiac MRI).

SECONDARY OUTCOMES:
Change in left ventricular function (E/e') | Baseline -18 months
  Measured average E/e' using Doppler-echocardiography
Change in left atrial volume index (LAV/BSA*) | Baseline - 9 months
  Measured using Doppler Echocardiography between baseline and 9 months. (*BSA calculated using the DuBois formula)
Change in left atrial function measured as total left atrial ejection fraction (LAEF) | Baseline -18 months
  Measured as total LAEF ((LAVmax - LAVmin)/LAVmax, by cardiac MRI
Change in left atrial function measured as left atrial stroke volume index | Baseline -18 months
  Measured as left atrial stroke volume index (LAVmax - LAVmin)/BSA (measured using Du Bois formula), or LAVimax-LAVimin by cardiac MRI
Change in left ventricular structure measured as LVMi | Baseline -18 months
  Measured using left ventricular mass index (LVMi), indexed to BSA (calculated using the DuBois formula) using cardiac MRI
Change in left ventricular function (LVEF) | Baseline -18 months
  Measured as left ventricular ejection fraction (LVEF) using cardiac MRI
Change in measures of vascular compliance (pulse pressure) | Baseline -18 months
  Measured using pulse pressure calculated from 24 hour ABPM measurements
Change in natriuretic peptide biomarker profile | Baseline -18 months
  Defined as log-transformed NT-proBNP
Time to first all cardiovascular death and major adverse cardiac events (MACE) requiring hospitalisation over 18 months | Baseline - 18 months
  MACE includes arrythmia (including atrial fibrillation/flutter), transient ischaemic attack, stroke, valvular heart disease, myocardial infarction, peripheral or pulmonary thrombosis/embolus or heart failure
Change in Left Atrial Volume Index (LAVi) analysed per protocol. | Baseline - 18 months
  Measured as left atrial volume (Simpson's method, using a stack of short axis slices across the entire left atrium) indexed to body surface area (DuBois formula) using Cardiac Magnetic Resonance Imaging (cardiac MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Ryan, Co-Investigator, PhD, Study Director — Heartbeat Trust, 3 Crofton Terrace, Dun Laoghaire, Co Dublin
Locations (2):
- Ireland (2):
  - The STOP-HF Service, St Michael's Hosptial, Dún Laoghaire, Co Dublin
  - St Vincents University Hospital, Dublin

REFERENCES:
- [Background] Ledwidge M, Gallagher J, Conlon C, Tallon E, O'Connell E, Dawkins I, Watson C, O'Hanlon R, Bermingham M, Patle A, Badabhagni MR, Murtagh G, Voon V, Tilson L, Barry M, McDonald L, Maurer B, McDonald K. Natriuretic peptide-based screening and collaborative care for heart failure: the STOP-HF randomized trial. JAMA. 2013 Jul 3;310(1):66-74. doi: 10.1001/jama.2013.7588. PMID 23821090
- [Background] Huelsmann M, Neuhold S, Resl M, Strunk G, Brath H, Francesconi C, Adlbrecht C, Prager R, Luger A, Pacher R, Clodi M. PONTIAC (NT-proBNP selected prevention of cardiac events in a population of diabetic patients without a history of cardiac disease): a prospective randomized controlled trial. J Am Coll Cardiol. 2013 Oct 8;62(15):1365-72. doi: 10.1016/j.jacc.2013.05.069. Epub 2013 Jun 27. PMID 23810874
- [Background] Phelan D, Watson C, Martos R, Collier P, Patle A, Donnelly S, Ledwidge M, Baugh J, McDonald K. Modest elevation in BNP in asymptomatic hypertensive patients reflects sub-clinical cardiac remodeling, inflammation and extracellular matrix changes. PLoS One. 2012;7(11):e49259. doi: 10.1371/journal.pone.0049259. Epub 2012 Nov 12. PMID 23152884
- [Background] Potter LR, Abbey-Hosch S, Dickey DM. Natriuretic peptides, their receptors, and cyclic guanosine monophosphate-dependent signaling functions. Endocr Rev. 2006 Feb;27(1):47-72. doi: 10.1210/er.2005-0014. Epub 2005 Nov 16. PMID 16291870
- [Background] Gardner DG, Chen S, Glenn DJ, Grigsby CL. Molecular biology of the natriuretic peptide system: implications for physiology and hypertension. Hypertension. 2007 Mar;49(3):419-26. doi: 10.1161/01.HYP.0000258532.07418.fa. Epub 2007 Feb 5. No abstract available. PMID 17283251
- [Background] Hogg K, Swedberg K, McMurray J. Heart failure with preserved left ventricular systolic function; epidemiology, clinical characteristics, and prognosis. J Am Coll Cardiol. 2004 Feb 4;43(3):317-27. doi: 10.1016/j.jacc.2003.07.046. PMID 15013109
- [Background] Querejeta R, Lopez B, Gonzalez A, Sanchez E, Larman M, Martinez Ubago JL, Diez J. Increased collagen type I synthesis in patients with heart failure of hypertensive origin: relation to myocardial fibrosis. Circulation. 2004 Sep 7;110(10):1263-8. doi: 10.1161/01.CIR.0000140973.60992.9A. Epub 2004 Aug 16. PMID 15313958
- [Background] Martos R, Baugh J, Ledwidge M, O'Loughlin C, Conlon C, Patle A, Donnelly SC, McDonald K. Diastolic heart failure: evidence of increased myocardial collagen turnover linked to diastolic dysfunction. Circulation. 2007 Feb 20;115(7):888-95. doi: 10.1161/CIRCULATIONAHA.106.638569. Epub 2007 Feb 5. PMID 17283265
- [Background] Ahmed SH, Clark LL, Pennington WR, Webb CS, Bonnema DD, Leonardi AH, McClure CD, Spinale FG, Zile MR. Matrix metalloproteinases/tissue inhibitors of metalloproteinases: relationship between changes in proteolytic determinants of matrix composition and structural, functional, and clinical manifestations of hypertensive heart disease. Circulation. 2006 May 2;113(17):2089-96. doi: 10.1161/CIRCULATIONAHA.105.573865. Epub 2006 Apr 24. PMID 16636176
- [Background] Nishikimi T, Maeda N, Matsuoka H. The role of natriuretic peptides in cardioprotection. Cardiovasc Res. 2006 Feb 1;69(2):318-28. doi: 10.1016/j.cardiores.2005.10.001. Epub 2005 Nov 10. PMID 16289003
- [Background] Solomon SD, Zile M, Pieske B, Voors A, Shah A, Kraigher-Krainer E, Shi V, Bransford T, Takeuchi M, Gong J, Lefkowitz M, Packer M, McMurray JJ; Prospective comparison of ARNI with ARB on Management Of heart failUre with preserved ejectioN fracTion (PARAMOUNT) Investigators. The angiotensin receptor neprilysin inhibitor LCZ696 in heart failure with preserved ejection fraction: a phase 2 double-blind randomised controlled trial. Lancet. 2012 Oct 20;380(9851):1387-95. doi: 10.1016/S0140-6736(12)61227-6. Epub 2012 Aug 26. PMID 22932717
- [Background] Watson CJ, Glezeva N, Horgan S, Gallagher J, Phelan D, McDonald K, Tolan M, Baugh J, Collier P, Ledwidge M. Atrial Tissue Pro-Fibrotic M2 Macrophage Marker CD163+, Gene Expression of Procollagen and B-Type Natriuretic Peptide. J Am Heart Assoc. 2020 Jun 2;9(11):e013416. doi: 10.1161/JAHA.119.013416. Epub 2020 May 20. PMID 32431194
- [Background] Januzzi JL Jr, Prescott MF, Butler J, Felker GM, Maisel AS, McCague K, Camacho A, Pina IL, Rocha RA, Shah AM, Williamson KM, Solomon SD; PROVE-HF Investigators. Association of Change in N-Terminal Pro-B-Type Natriuretic Peptide Following Initiation of Sacubitril-Valsartan Treatment With Cardiac Structure and Function in Patients With Heart Failure With Reduced Ejection Fraction. JAMA. 2019 Sep 17;322(11):1085-1095. doi: 10.1001/jama.2019.12821. PMID 31475295
- [Background] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Background] Ibrahim NE, McCarthy CP, Shrestha S, Gaggin HK, Mukai R, Szymonifka J, Apple FS, Burnett JC Jr, Iyer S, Januzzi JL Jr. Effect of Neprilysin Inhibition on Various Natriuretic Peptide Assays. J Am Coll Cardiol. 2019 Mar 26;73(11):1273-1284. doi: 10.1016/j.jacc.2018.12.063. PMID 30898202
- [Background] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Derived] Ledwidge M, Dodd JD, Ryan F, Sweeney C, McDonald K, Fox R, Shorten E, Zhou S, Watson C, Gallagher J, McVeigh N, Murphy DJ, McDonald K. Effect of Sacubitril/Valsartan vs Valsartan on Left Atrial Volume in Patients With Pre-Heart Failure With Preserved Ejection Fraction: The PARABLE Randomized Clinical Trial. JAMA Cardiol. 2023 Apr 1;8(4):366-375. doi: 10.1001/jamacardio.2023.0065. PMID 36884247

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04687111/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT04687111/ICF_000.pdf